CLINICAL TRIAL: NCT07165860
Title: Novel Doula Intervention to Leverage Clinic-community Connections to Support Perinatal Intimate Partner Violence Survivors
Brief Title: Clinical Trial to Reduce Perinatal Intimate Partner Violence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Maya Ragavan, Associate Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY24080042; R01NR021484 (NIH)
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Domestic Violence; Perinatal Problems
Keywords: intimate partner violence; perinatal health; doula
MeSH Terms: interventions — Doulas; Nicotine

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The trial will be blinded to the investigators and participants will be unblinded if a participant is experiencing distress or needs support from the primary investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active control arm (Active Comparator): The active control arm will include two structured check-ins by a trained intimate partner violence advocate from a local victim services agency. The IPV advocate will check in twice: once prenatally (after randomization) and the next postpartum. All participants in the active control arm will have access to the 24/7 helpline.
  Interventions: Behavioral: Thrive
- Doula group (intervention) (Experimental): The intervention arm will include support rom a community-based doula connected with an IPV survivor during the second trimester and followed for 6 months. The doulas will provide full-spectrum services, which include attending clinic visits, support during the delivery, telephone and virtual check-ins, and connection to resources. Doulas have 4 structured visits (4 hours) and the rest of the time will be unstructured. Doulas will also attend the participant's birth. Doulas will provide a trauma-informed perinatal workbook to the participants that our team developed.
  Interventions: Behavioral: Doulas

INTERVENTIONS:
Behavioral: Doulas — The intervention will be pairing intimate partner violence survivors with a trained doula
  Arms: Doula group (intervention)
Behavioral: Thrive — The active control arm will include pairing intimate partner violence survivors with IPV advocates
  Arms: Active control arm

SUMMARY:
This is a two-armed, fully powered hybrid type 1 trial to test the effectiveness of a doula intervention compared with an active control in reducing intimate partner violence (IPV) among perinatal IPV survivors

DETAILED DESCRIPTION:
The study team will complete a 2-arm randomized clinical trial to test the effectiveness of IPV-trained doulas compared with an active control in reducing IPV among perinatal IPV survivors. Participants randomized into doula group will be paired community doula who will provide full-spectrum doula services prenatally (22 weeks gestation), through the birthing period, to early postpartum (6 months total). Participants randomized to the active two structured intakes from a victim services agency. Participants will be recruited from their prenatal visit at 1 of 3 sites with 163 perinatal people randomized to the doula group and 163 randomized to active control (N=326). The primary outcome is change in IPV across a range coercive behaviors from baseline to 12-months post enrollment. Secondary outcomes include change in cannabis and tobacco use, as well as depressive symptoms, anxiety, and unmet basic needs. The study will also be assessing changes in intermediate outcomes, including resource utilization, trust of doulas and IPV advocates, parenting stress, safety-related empowerment, and social support. Measures will be completed at enrollment, and then 3-, 6-, and 12-months post-enrollment. In Aim 2, the study team will be assessing potential mediators and moderators driving intervention effects and in Aim 3, collecting information about implementation outcomes.

ELIGIBILITY:
Inclusion Criteria: Perinatal IPV survivors are eligible if they:

* 1) feel comfortable completing the study in Spanish or English
* 2) are age 18 or older
* 3) are no more than 22 weeks gestation
* 4) identify as an IPV survivor by answering affirmatively to a definition of experiencing IPV
* 5) live within a 50 mile radius of Pittsburgh, Pennsylvania
* 6) able to provide safe and complete contact information or take a study cell phone

Exclusion Criteria:

* Unable to consent
* Do not meet inclusion criteria
* Cannot provide safe contact information or take a study cell phone
* Incarcerated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Perinatal physical, sexual, or emotional abuse (past 3 months) | baseline, 3 months, 6 months, 12 months
  15 item Composite Abuse Scale Short form, scale is 0 to 5 and 15 items are added for a summary score, higher number means more IPV
Substance use coercion (past 3 month) | baseline, 3 months, 6 months, and 12 months
  5 item measure answer choices and yes/no
Mental health coercion (past 3 month) | baseline, 3 months, 6 months, and 12 months
  5 item mental health coercion survey with yes and no answer choices
Economic Abuse (past 3 month) | baseline, 3 month, 6 months, and 12 months
  12 item Revised Scale of Economic Abuse (answer choices yes or no), more yes responses means more experiences of economic abuse
Reproductive Coercion (past 3 months) | baseline, 3 months, 6 months, and 12 months
  9 item reproductive coercion scale (answer choices yes/no). More yes responses means more experiences of reproductive coercion
Sleep coercion (past 3 months) | baseline, 3 months, 6 months, and 12 months
  1 item sleep coercion measure (investigator developed, yes/no)

SECONDARY OUTCOMES:
Substance use | baseline
  4 item validated measure to assess substance use during pregnancy
Tobacco use | baseline, 3 months, 6 months, 12 months
  Type, frequency, use currently and before pregnancy (4 items)
Depressive symptoms | baseline, 3 months, 6 months, 12 months
  10 item Edinburgh Postnatal Depression Scale; α=0.87, summary scale and mean, higher score means more depression. Scale ranges from 0 to 30
Anxiety | baseline, 3 months, 6 months, and 12 months
  7 item validated GAD-7, scores Likert 0 to 3, added up for summary scale, higher score means more anxiety. Scale ranges from 0 to 21
Unmet basic needs (financial, food, and housing insecurity) | Baseline, 12 months
  5 item investigator developed scale on food, housing, and utilities insecurity. Answer choices yes or no, more yes choices chosen means more unmet basic needs
Past 3-month substance use | 6 months, 12 months
  Substances used in the past 3 months, first yes/no and then type of substance

OTHER OUTCOMES:
Resource utilization | baseline, 3 months, 6 months, 12 months
  21 items; investigator developed examining utilization of local and national community-based resources; answer choices are yes and no
Safety related empowerment | baseline, 3 months, 6 months, 12 months
  13 item Measures of Victim Empowerment Related to Safety survey; α=0.87, answer choices 0 to 4, summary score created, higher score means more empowerment
Trust of healthcare, doula and IPV advocate | baseline, 3 months, 6 months, 12 months
  3 item investigator developed, answer choices 0 to 4. Each item analyzed separately (doula, IPV advocate, and physician)
Social support | baseline, 3 months, 6 months, 12 months
  12 item Multidimensional Scale of Perceived Social Support; α=0.93. Likert scale 1 to 7, summary score created, higher score means more feelings of social support
Everyday Discrimination | baseline and 12 months
  9-item Everyday Discrimination Scale; α=0.84. Answers scores on Likert scale, 0 to 5, summary score created, higher score means more experiences of discrimination. Scale ranges from 10 to 60
Major discrimination | baseline and 12 months
  9 item scale on experiences of major discrimination, answer choices yes or no, more yes answer choices means more experiences of major discrimination
Sleep coercion (lifetime) | baseline
  1 item sleep coercion measure (investigator developed, yes/no)
Reproductive Coercion (lifetime) | baseline
  9 item reproductive coercion scale (answer choices yes/no). More yes responses means more experiences of reproductive coercion
Economic Abuse (lifetime) | baseline
  12 item Revised Scale of Economic Abuse (answer choices yes or no), more yes responses means more experiences of economic abuse
Mental health coercion (lifetime) | baseline
  5 item mental health coercion survey with yes and no answer choices
Lifetime substance use coercion | baseline
  5 item measure answer choices and yes/no
Lifetime physical, sexual, or emotional abuse | baseline
  15 item Composite Abuse Scale Short form, scale is 0 to 5 and 15 items are added for a summary score, higher number means more IPV
Self-efficacy | baseline, 3, 6 and 12 months
  Validated 8 item New General Self Efficacy Scale. Likert scale 1 to 5, summary scale created, a higher score means more self-efficacy. The score ranges from 10 to 40
Parenting Stress | 6 months, 12 months
  Validated Parenting Stress Scale; 18 items; Likert Scale 1 to 5, summary score created, a higher score means more parenting stress. The range is 18 to 90

CONTACTS AND LOCATIONS:
Overall Officials: Maya I Ragavan, Principal Investigator — University of Pittsburgh; Dara Mendez, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - The Midwife Center, Pittsburgh, Pennsylvania
  - Family Medicine Department, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No individual level data will be shared outside of our team. Aggregated data may be shared.